CLINICAL TRIAL: NCT05991323
Title: A Prospective Observational Study of Patients Receiving Dupilumab for Prurigo Nodularis
Brief Title: Real-World Effectiveness of Dupilumab in Patients With Prurigo Nodularis: An Observational Study
Acronym: GLOBOSPIN
Status: Active, not recruiting | Type: Observational
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: OBS17721; U1111-1288-8567 (Registry Identifier: ICTRP)
Record Dates: First submitted 2023-07-19; First posted 2023-08-14 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Prurigo Nodularis
MeSH Terms: interventions — dupilumab

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient with prurigo nodularis: Participants aged 18 years or older who start receiving dupilumab for prurigo nodularis (according to the country-specific prescribing information) prior to and independently of their participation in the study
  Interventions: Drug: Dupilumab

INTERVENTIONS:
Drug: Dupilumab — Injection solution; subcutaneous
  Other Names: DUPIXENT; SAR231893

SUMMARY:
This study is a prospective, multinational, observational investigation designed to elucidate the real-world effectiveness and treatment patterns of dupilumab therapy in adult patients diagnosed with prurigo nodularis (PN).

The primary objective of this study is to comprehensively characterize the real-world usage of dupilumab for the management of PN.

In addition to this, the study aims to achieve several secondary objectives, including a detailed assessment of the medical history, socio-demographic and disease characteristics of dupilumab-treated PN patients, as well as the evaluation of the long-term real-world effectiveness of dupilumab therapy for PN.

DETAILED DESCRIPTION:
The follow-up period will be 18 months or until death, loss to follow-up, or withdrawal, whichever comes first.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older at the time of informed consent.
* Physician decision to treat the patient with dupilumab for prurigo nodularis (according to the country-specific prescribing information) made prior to and independently of the patient's participation in the study.
* Patients able to understand and complete study-related questionnaires.
* Patients provide voluntary informed consent to participate in the study before inclusion in the study.

Exclusion Criteria:

* Patients who have a contraindication to dupilumab according to the country-specific prescribing information label.
* Any condition that, in the opinion of the Investigator, may interfere with the patient's ability to participate in the study, such as short life expectancy, substance abuse, severe cognitive impairment, or other comorbidities that can predictably prevent the patient from completing the schedule of visits and assessments.
* Patients currently participating in any interventional clinical trial.
* Prior use of dupilumab within 6 months of the screening visit, or within 6 months of the baseline visit if screening and baseline occur on the same day.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible participants who initiate dupilumab treatment for prurigo nodularis (according to the country-specific prescribing information)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-12-12 (Actual); Primary Completion 2026-09-22 (Estimated); Study Completion 2026-09-22 (Estimated)

PRIMARY OUTCOMES:
Frequency of reasons for dupilumab treatment initiation with the description of dosing, frequency and duration of treatment | At baseline
Frequency of reasons for dupilumab treatment modifications with the description of the modified treatment | From baseline up to month 18
Proportion of patients who discontinued dupilumab | From baseline up to month 18
Frequency of reasons for dupilumab treatment discontinuation | From baseline up to month 18
Proportion of patients hospitalized due to PN | From baseline up to month 18

SECONDARY OUTCOMES:
Baseline Characteristics: PN-related medical history | At baseline
  (e.g., date of diagnosis, severity, comorbidities)
Baseline Characteristics: Socio-demographics of PN patients | At baseline
  (e.g., month and year of birth (where allowed) or age, gender, race (if allowed), ethnicity (if allowed), Fitzpatrick skin type)
Baseline Characteristics: Type of PN therapies received prior to initiation of dupilumab treatment | At baseline
Proportion of patients using concomitant medication | At baseline
Proportion of patients with a ≥ four-point improvement (reduction) in Worst Itch Numeric Rating Scale (WI-NRS) | From baseline up to month 18
  The WI-NRS is a single-item Patient-Reported Outcomes (PRO). Patients will be asked to report the intensity of their worst pruritus (itch) using the 0 to 10 WI-NRS. Scores range from 0 to 10, with higher scores indicating greater itch intensity.
Mean change in WI-NRS | From baseline up to month 18
  The WI-NRS is a single-item Patient-Reported Outcomes (PRO). Patients will be asked to report the intensity of their worst pruritus (itch) using the 0 to 10 WI-NRS. Scores range from 0 to 10, with higher scores indicating greater itch intensity.
Proportion of patients with a ≥ four-point improvement (reduction) in Skin Pain Numeric Rating Scale (NRS) | From baseline up to month 18
  The Skin Pain NRS is a single-item Patient-Reported Outcomes (PRO). Patients indicate the intensity of their worst skin pain over the past 24 hours by selecting a number on the scale that ranges from 0 ("No pain") to 10 ("Worst pain imaginable"). Scores range from 0 to10, with higher scores indicating greater pain intensity.
Mean change in Skin Pain NRS | From baseline up to month 18
  The Skin Pain NRS is a single-item Patient-Reported Outcomes (PRO). Patients indicate the intensity of their worst skin pain over the past 24 hours by selecting a number on the scale that ranges from 0 ("No pain") to 10 ("Worst pain imaginable"). Scores range from 0 to10, with higher scores indicating greater pain intensity.
Proportion of patients with a ≥ two-point improvement (reduction) in Sleep Disturbance Numeric Rating Scale (NRS) | From baseline up to month 18
  The Sleep Disturbance NRS is a single-item Patient-Reported Outcomes (PRO). Patients will be asked to report the severity of their sleep disturbance using a 0 to 10 NRS. Scores range from 0 to10, with higher scores indicating worse sleep quality.
Mean change in Sleep Disturbance NRS | From baseline up to month 18
  The Sleep Disturbance NRS is a single-item Patient-Reported Outcomes (PRO). Patients will be asked to report the severity of their sleep disturbance using a 0 to 10 NRS. Scores range from 0 to10, with higher scores indicating worse sleep quality.
Proportion of patients with Patient Global Impression of Change of PN Disease (PGIC) score of "Very much better (improved)" | From baseline up to month 18
  The PGIC is a 7-point scale to assess patient health and determine if there has been an improvement or decline in clinical status. Scores range from 1 to 7, with higher score indicating worse health status.
Proportion of patients with PGIC score of "Very much better (improved)" or "Moderately better (improved)" | From baseline up to month 18
  The PGIC is a 7-point scale to assess patient health and determine if there has been an improvement or decline in clinical status. Scores range from 1 to 7, with higher score indicating worse health status.
Mean change in PGIC | From baseline up to month 18
  The PGIC is a 7-point scale to assess patient health and determine if there has been an improvement or decline in clinical status. Scores range from 1 to 7, with higher score indicating worse health status.
Proportion of patients with Patient Global Impression of Severity of PN Disease (PGIS) score of "None" | From baseline up to month 18
  The PGIS is a one-item questionnaire that asks participants to provide the overall self-assessment of their disease severity on a 4-point scale for the past week. Scores range from 1 to 4, with higher score indicating worse symptom severity.
Proportion of patients with PGIS score of "None" or "Mild" | From baseline up to month 18
  The PGIS is a one-item questionnaire that asks participants to provide the overall self-assessment of their disease severity on a 4-point scale for the past week. Scores range from 1 to 4, with higher score indicating worse symptom severity.
Mean change in PGIS | From baseline up to month 18
  The PGIS is a one-item questionnaire that asks participants to provide the overall self-assessment of their disease severity on a 4-point scale for the past week. Scores range from 1 to 4, with higher score indicating worse symptom severity.
Mean change in Dermatology Life Quality Index (DLQI) | From baseline up to month 18
  The DLQI is designed to measure the health-related quality of life of adults with a skin disease. The DLQI consists of 10 questions related to the effect of skin disease over the past week. Overall scoring ranges from 0 to 30, with a high score indicative of a poorer Health-Related Quality of Life (HRQoL)
Mean change in Pruritus Activity Score (PAS) | From baseline up to month 18
  The modified PAS is a clinical-reported measure that evaluates the pruritic lesions. The modified questionnaire consists of five items: the type (visible lesions: item 1a; predominant lesions: item1b), estimated number (item 2), distribution (item 3), the representative body area and exact number of lesions (item 4), and the activity in terms of percentage of pruriginous lesions with excoriations/crusts on top (reflecting active scratching; item 5a) and the percentage of healed pruriginous lesions (reflecting healing of chronic prurigo; item 5b). The modified PAS will be completed based on the standard of care clinical assessment.
Proportion of patients with Investigator's Global Assessment-chronic prurigo Activity (IGA-CPG Activity) score of 0 or 1 | From baseline up to month 18
  The IGA-CPG Activity is an instrument used to assess the overall activity of chronic prurigo lesions at a given time point, as determined by the Investigator. In this context, nodules, papules, plaques and other PN related lesions are defined as pruriginous lesions or chronic prurigo lesions. The instrument consists of a five-point scale ranging from 0 to 4. Higher scores indicate severe CPG.
Mean change in IGA-CPG Activity | From baseline up to month 18
  The IGA-CPG Activity is an instrument used to assess the overall activity of chronic prurigo lesions at a given time point, as determined by the Investigator. In this context, nodules, papules, plaques and other PN related lesions are defined as pruriginous lesions or chronic prurigo lesions. The instrument consists of a five-point scale ranging from 0 to 4. Higher scores indicate severe CPG.
Proportion of patients with Investigator's Global Assessment-chronic prurigo Stage (IGA-CPG Stage) score of 0 or 1 | From baseline up to month 18
  The IGA-CPG Stage is an instrument used to assess the overall number and thickness of chronic prurigo lesions at a given time point, as determined by the Investigator. In this context, nodules, papules, plaques and other PN related lesions are defined as pruriginous lesions or chronic prurigo lesions. The instrument consists of a five-point scale ranging from 0 to 4. Higher scores indicate severe CPG.
Mean change in IGA-CPG Stage | From baseline up to month 18
  The IGA-CPG Stage is an instrument used to assess the overall number and thickness of chronic prurigo lesions at a given time point, as determined by the Investigator. In this context, nodules, papules, plaques and other PN related lesions are defined as pruriginous lesions or chronic prurigo lesions. The instrument consists of a five-point scale ranging from 0 to 4. Higher scores indicate severe CPG.
Mean change in EQ-5D-5L | From baseline up to month 18
  The EQ-5D-5L comprises of five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. The patient is asked to indicate their health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
Mean change in Hospital Anxiety and Depression Scale (HADS) total score | From baseline up to month 18
  The HADS is a Patient-Reported Outcomes (PRO) instrument for screening anxiety and depression in non-psychiatric populations. The HADS consists of 14 items, 7 each for anxiety and depression symptoms. Patients select a response from 0 to 3 for each item, based on how they have been feeling in the past week. Scores range from 0 to 21 for each subscale. HADS anxiety (HADS-A) and HADS depression (HADS-D) scores ≤ 7 indicate no clinically relevant symptoms (normal), 8 to 10 borderline abnormal (borderline case), and 11 to 21 abnormal (maximum 21) indicating more severe symptoms.
Proportion of patients reported working, absenteeism score, presenteeism score, and overall impairment working score using the Work Productivity and Activity Impairment (WPAI) questionnaire | From baseline up to month 18
  The Work Productivity and Activity Impairment General Health (WPAI-GH) is a 6-item Patient-Reported Outcomes (PRO) instrument that measures the effect of a condition on productivity during work and regular activities in the seven days prior to completion. The instrument comprises 4 domains: absenteeism, presenteeism, overall work impairment, and activity impairment due to health. WPAI-GH outcomes are expressed as impairment percentages, with higher numbers indicating greater impairment and less productivity, i.e., worse outcomes.
Percentage of patients experiencing AEs and SAEs | From baseline up to month 18

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (49):
- United States (23):
  - Medical Dermatology Specialists Site Number : 8400005, Phoenix, Arizona
  - Saguaro Dermatology Associates, LLC - Probity - PPDS- Site Number : 8400024, Phoenix, Arizona
  - Center for Dermatology Clinical Research- Site Number : 8400002, Fremont, California
  - Halcyon Dermatology- Site Number : 8400023, Laguna Hills, California
  - Mission Dermatology - Rancho Santa Margarita- Site Number : 8400015, Rancho Santa Margarita, California
  - Golden State Dermatology- Site Number : 8400014, Walnut Creek, California
  - Total Vein And Skin, LLC- Site Number : 8400019, Boynton Beach, Florida
  - GSI Clinical Research- Site Number : 8400017, Margate, Florida
  - Allergy Center at Brookstone Research - Centricity Research - PPDS- Site Number : 8400025, Columbus, Georgia
  - Dawes Fretzin Clinical Research Group-7910 N Shadeland Ave- Site Number : 8400003, Indianapolis, Indiana
  - Oakland Hills Dermatology - 3400 Auburn Rd- Site Number : 8400007, Auburn Hills, Michigan
  - Derm Institute of Western Michigan- Site Number : 8400034, Caledonia, Michigan
  - Dermatology Associates Western Michigan- Site Number : 8400033, Grand Rapids, Michigan
  - U.S. Dermatology Partners Lee's Summit- Site Number : 8400016, Lee's Summit, Missouri
  - University of Nebraska - Lauritzen Outpatient Center- Site Number : 8400029, Omaha, Nebraska
  - Vivida Dermatology - Flamingo- Site Number : 8400013, Las Vegas, Nevada
  - Las Vegas Dermatology- Site Number : 8400027, Las Vegas, Nevada
  - Duke Dermatology Clinic- Site Number : 8400026, Durham, North Carolina
  - Medical University of South Carolina (MUSC) - PPDS- Site Number : 8400001, Charleston, South Carolina
  - North Texas Center for Clinical Research- Site Number : 8400012, Frisco, Texas
  - U.S. Dermatology Partners Longview- Site Number : 8400032, Longview, Texas
  - Texas Tech University Health Sciences Center-125 W Hague Rd- Site Number : 8400010, Lubbock, Texas
  - West Virginia Research Institute- Site Number : 8400030, Morgantown, West Virginia
- Canada (10):
  - Investigational Site Number : 1240009, Calgary, Alberta
  - Investigational Site Number : 1240007, Edmonton, Alberta
  - Investigational Site Number : 1240012, Surrey, British Columbia
  - Investigational Site Number : 1240006, Fredericton, New Brunswick
  - Investigational Site Number : 1240004, Ajax, Ontario
  - Investigational Site Number : 1240003, Barrie, Ontario
  - Investigational Site Number : 1240011, London, Ontario
  - Investigational Site Number : 1240002, Newmarket, Ontario
  - Investigational Site Number : 1240005, Toronto, Ontario
  - Investigational Site Number : 1240010, Waterloo, Ontario
- China (9):
  - Investigational Site Number : 1560009, Guangzhou, Guangdong
  - Investigational Site Number : 1560004, Xi'an, Shaanxi
  - Investigational Site Number : 1560003, Jinan, Shandong
  - Investigational Site Number : 1560008, Hangzhou, Zhejiang
  - Investigational Site Number : 1560010, Wenzhou, Zhejiang
  - Investigational Site Number : 1560007, Beijing
  - Investigational Site Number : 1560005, Beijing
  - Investigational Site Number : 1560006, Shanghai
  - Investigational Site Number : 1560002, Shenzhen
- France (2):
  - Investigational Site Number : 2500005, Brest, Finistère
  - Investigational Site Number : 2500001, Nantes
- Japan (3):
  - Investigational Site Number : 3920001, Obihiro, Hokkaido
  - Investigational Site Number : 3920003, Kyoto
  - Investigational Site Number : 3920004, Matsudo
- Netherlands (2):
  - Investigational Site Number : 5280001, Bergen op Zoom, North Brabant
  - Investigational Site Number : 5280002, Hoofddorp, North Holland

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org